CLINICAL TRIAL: NCT02068157
Title: Interstitial Photodynamic Therapy During Standard Chemotherapy for Palliation of Patients With Head and Neck Squamous Cell Carcinoma - Phase II
Brief Title: Interstitial Photodynamic Therapy in Treating Patients With Recurrent Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study no longer has an active IDE
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 235613; NCI-2014-00210 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 235613 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2014-02-18; First posted 2014-02-21 (Estimated); Results first posted 2017-08-28 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-09

CONDITIONS: Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Laryngeal Verrucous Carcinoma; Recurrent Lip and Oral Cavity Squamous Cell Carcinoma; Recurrent Metastatic Squamous Cell Carcinoma in the Neck With Occult Primary; Recurrent Oral Cavity Verrucous Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Tongue Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lymphoid Interstitial Pneumonia; Tongue Neoplasms | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Phototherapy; Dihematoporphyrin Ether; Trioxsalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (porfimer sodium, image-guided I-PDT) (Experimental): Patients receive porfimer sodium IV over 3-5 minutes on day 0. Patients then undergo image-guided I-PDT on day 2.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Photodynamic Therapy; Drug: Porfimer Sodium

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Photodynamic Therapy — Undergo image-guided I-PDT
  Other Names: PDT; Photoradiation Therapy
Drug: Porfimer Sodium — Given IV
  Other Names: CL-184116; DHE; Dihematoporphyrin Ester; Dihematoporphyrin Ether; Photofrin II

SUMMARY:
This phase II trial studies the effects of interstitial photodynamic therapy in patients with head and neck cancer that has come back. Interstitial photodynamic therapy uses a combination of laser light and a light-sensitive drug called porfimer sodium to destroy tumors. During treatment a laser light is used to activate the drug. Interstitial photodynamic therapy may be an effective treatment for head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate that our image-guided interstitial photodynamic therapy (I-PDT) dosimetry system can be used to tailor this therapy to individual patients.

OUTLINE:

Patients receive porfimer sodium intravenously (IV) over 3-5 minutes on day 0. Patients then undergo image-guided I-PDT on day 2.

After completion of study, patients are followed up at 1 month, 2 months, 4 months, and then every 2 months for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Histologically confirmed recurrent squamous cell carcinoma of the oral cavity, pharynx, (oropharynx, larynx) and neck
* Tumor accessible for unrestricted illumination for interstitial photodynamic therapy (PDT) (accessibility as determined by the physician)
* Patients on chemotherapy &/or targeted agents for palliation
* Life expectancy of at least 6 months in the judgment of the physician
* Subjects of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for 6 months after the last treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Subject or legal representative must understand the investigational nature of this study and sign an Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Radiotherapy within the last 2 months in the area to be treated
* Patients with known brain metastases should be excluded from this clinical trial
* Tumor invading a major blood vessel (such as the carotid artery)
* Tumor is not clearly shown on a computed tomography (CT) scan
* Location and extension of the tumor precludes an effective I-PDT
* Patients with porphyria, or with known hypersensitivity to porphyrins or porphyrin-like compounds
* While blood cell (WBC) < 2.0 x 10^9/L
* Total serum bilirubin > 2.0 mg/dl
* Serum creatinine > 2 mg/dl
* Alkaline phosphatase (hepatic) > 3 times the upper normal limit
* Serum glutamic oxaloacetic transaminase (SGOT) > 3 times the upper limit of normal
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, acute exacerbation of congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or nursing female subjects
* Unwilling or unable to follow protocol requirements and the light exposure precautions
* Any condition which in the Investigators' opinion deems the subject an unsuitable candidate to receive study drug and therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2016-10-13 (Actual); Study Completion 2016-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Arshad, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Porfimer Sodium, Image-guided I-PDT)
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Treatment (Porfimer Sodium, Image-guided I-PDT)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response or Partial Response According to RECIST v1.1
Description: Tumor response rate according to Response Evaluation Criteria in Solid Tumors 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 12 months
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Porfimer Sodium, Image-guided I-PDT)
Number analyzed (Participants) | 3
percentage of participants | 33 [1 to 91]

2. Secondary Outcome: Serum Alkaline DNase (SADA) Activity
Description: SADA activity will be correlated with tumor response according to the guidelines of the revised Response Criteria in Solid Tumors 1.1.
Time Frame: Up to 12 months
Population: The published assay could not be validated in murine samples. As such, no human samples were analyzed.
Arm/Group | Treatment (Porfimer Sodium, Image-guided I-PDT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Porfimer Sodium, Image-guided I-PDT)
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Porfimer Sodium, Image-guided I-PDT) (N=3)
Pain (General disorders) | 1 (35)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Porfimer Sodium, Image-guided I-PDT) (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (23)
Ear pain (Ear and labyrinth disorders) | 1 (9)
Eye irritation (Eye disorders) | 1 (6)
Eye swelling (Eye disorders) | 1 (5)
Fatigue (General disorders) | 1 (26)
Injection site pain (General disorders) | 1 (9)
Sunburn (Injury, poisoning and procedural complications) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (10)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (23)
Rash (Skin and subcutaneous tissue disorders) | 1 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes